CLINICAL TRIAL: NCT04885556
Title: Evaluation of a Novel Female Hygiene Device for Postcoital Discomfort
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, Michael Ingber, Director of The Center for Specialized Women's Health, division of Garden State Urology/Atlantic Health System, Atlantic Health System
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC-004
Record Dates: First submitted 2021-04-28; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Vaginal Discharge; Dyspareunia; Female Sexual Dysfunction; Vaginitis; Bacterial Vaginoses
Keywords: vaginal discharge; dripping; vaginal odor
MeSH Terms: conditions — Vaginal Discharge; Dyspareunia; Vaginitis; Vaginosis, Bacterial

STUDY DESIGN:
Intervention Model Description: Subjects to be placed into one of two study groups, 1) immediate use and 2) 1 hour use
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Immediate Use (Experimental): Subjects in this arm will be instructed to use the study device for 2 minutes and remove
  Interventions: Device: Tampon-like device for absorption of sexual fluids
- 1 hour use (Experimental): Subjects in this arm will be instructed to use the product for one hour and then remove
  Interventions: Device: Tampon-like device for absorption of sexual fluids

INTERVENTIONS:
Device: Tampon-like device for absorption of sexual fluids — Subjects will insert a tampon-like device to absorb sexual fluids after intercourse

SUMMARY:
Previous research has shown that semen deposition in the vagina after intercourse leads to dripping, discomfort, and vaginal odor. This study is evaluating a hygiene device designed to be inserted into the vagina after intercourse to absorb semen deposited into the vaginal canal to determine if there is a reduction in dripping and odor, and to determine the amount of fluids absorbed.

DETAILED DESCRIPTION:
Despite the significant number of sexual dysfunctions in women, physicians often avoid discussing these concerns in the office setting. With recent research on the role of the pelvic floor, and recently approved medical therapies for hypoactive sexual desire disorder, physicians have begun to adapt to questioning patients about libido and pain-related sexual dysfunctions. However, pain-related sexual questionnaires often focus on insertional and penetrational dyspareunia, without asking about discomfort minutes, hours, or even the day following sexual intercourse. One common compliant in ambulatory sexual medicine clinics is the bothersome dripping, odor, and discomfort women experience after sexual activity when no condom is used, and when intravaginal ejaculation occurs.

Previous studies have shown the effects of semen on alterations in the vaginal flora. These changes contribute to a multitude of clinical complaints and diagnoses, including malodor, continuous discharge after intercourse, and bacterial vaginosis (BV). The exposure of semen changes the vaginal flora by increasing the pH levels, in turn altering the bacterial growth pattern. This implies the persistent presence of semen in the vagina may be one of the causes of malodor and development of BV. Chvapil utilized gas chromatography and demonstrated that the longer period of time semen was present in the vagina, the more likely it resulted in a strong and unattractive vaginal odor. Gallo showed that an incidental diagnosis of BV was correlated with detection of sperm on gram stain, and frequent coitus with or without condom use.

The investigator's goal in this study is to evaluate a novel postcoital consumer health product and its effects on the complaints of continuous seepage of semen and vaginal odor after intercourse.

ELIGIBILITY:
Inclusion Criteria:

* Heterosexual
* Age 25-50
* Has used tampons in the past 5 years
* Sexually active (vaginal intercourse, minimum once per week)
* Answered "moderate" to "severe" to being bothered by dripping/discomfort on Patient Global Impression of Severity (PGI-S) questionnaire "on minutes, hours, or following day"
* Willing and able to use product
* Understands, reads, writes, and speaks English

Exclusion Criteria:

* Pregnant
* Currently using condoms
* Unable to use device due to poor motor function
* Chronic disease which makes prone to infection (diabetes, autoimmune)
* Recurrent yeast infections
* Recurrent Urinary tract infection (UTI) (>2 within the past year)
* Diagnosis of pelvic organ prolapse (Stage II or greater)
* Previous pelvic or vaginal surgery which, in the opinion of the investigator, may prevent proper use of product
* Unable to sign informed consent

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-05 (Actual); Primary Completion 2021-09-15 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
Patient Global Impression of Improvement (PGI-I) | within 1 hour of use of product
  Validated Questionnaire
Weight of Investigational Device | within 1 hour of use of product
  Product weight (amount of fluid absorbed)

CONTACTS AND LOCATIONS:
Locations (1):
- The Center for Specialized Women's Health, division of Garden State Urology, Denville, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No